CLINICAL TRIAL: NCT00556400
Title: Treatment of Menorrhagia in Women With Thrombocytopenia: Comparison of Platelet Transfusion Alone to Platelet Transfusion With Continuous Oral Contraceptive Pills
Brief Title: Treatment of Menorrhagia in Women With Thrombocytopenia Using Platelets or Platelets and Hormones
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early termination because of insufficient accrual.
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 080022; 08-CH-0022 (Other: NIH Clinical Center protocol number)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Aplastic Anemia; Menorrhagia; Amenorrhea
Keywords: Uterine Bleeding; Thrombocytopenia; Aplastic Anemia; Oral Contraceptive Pills; Menorrhagia
MeSH Terms: conditions — Anemia, Aplastic; Menorrhagia; Amenorrhea; Uterine Hemorrhage; Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lo-ovral (Active Comparator): 1 tablet of lo-ovral is administered twice a day
  Interventions: Drug: Lo-Ovral Oral Contraceptive Pills
- sugar pill (Placebo Comparator): Sugar pill was provided as a placebo
  Interventions: Drug: Placebo - sugar pill

INTERVENTIONS:
Drug: Lo-Ovral Oral Contraceptive Pills
  Arms: Lo-ovral
Drug: Placebo - sugar pill
  Arms: sugar pill

SUMMARY:
This study will explore the role of oral contraceptive pills in managing uterine bleeding in women who have low blood platelet counts as a result of aplastic anemia. Oral contraceptive pills have been shown to be effective in managing uterine bleeding in healthy women, but the effects have not been thoroughly studied in women who have low platelet counts. The purpose of the study is to determine whether oral contraceptive pills are a useful complement to platelet transfusions in women with aplastic anemia and uterine bleeding.

Volunteers for this study must be women between 12 and 55 years of age who have been diagnosed with aplastic anemia (with a platelet count of less than 50,000/microliter) and currently have active uterine bleeding. Candidates must not be pregnant or breastfeeding, must have a uterus and at least one functioning ovary, and must be willing to use nonhormonal methods of birth control (such as condoms or a diaphragm) for the duration of the study. On the first visit, candidates will be screened with a complete medical history (including obstetric and gynecological history) and will undergo a physical examination, a pelvic exam and a pelvic ultrasound. Blood and urine samples will also be taken on this first visit.

The study will last approximately two weeks. Participants will be asked to monitor their medication doses and severity of bleeding during the course of the study. After the first visit, participants will be separated into two randomized groups and will receive either one tablet of oral contraceptive or a placebo twice daily, to be taken 12 hours apart at the same times each day. Participants will also receive platelet transfusions as needed to ensure that their platelet counts remain over 20,000/microliter. After seven days, researchers will assess participants' uterine bleeding and all participants will be given oral contraceptives in the second week of the study. Participants whose bleeding has decreased will receive only one tablet; participants who still have moderate to severe uterine bleeding will receive two tablets. A final assessment will be performed on day 14 of the study.

DETAILED DESCRIPTION:
Low platelet counts can occur as a result of blood diseases like bone marrow failure, or from undergoing procedures such as chemotherapy treatment or stem cell transplantation. A major complication of low platelet counts in reproductive aged women is uterine bleeding, which can be life threatening. Sometimes this bleeding begins with a normal menstrual cycle but may start unexpectedly. In either instance, stopping uterine bleeding not only requires blood products including platelets but also hormonal treatments.

The hormones estrogen or progesterone can aid in this setting presumably by promoting endometrial angiogenesis. Continuous oral contraceptive pills (OCP) have been shown to be very effective in the management of heavy menstrual bleeding in healthy women, but few studies have been carried out in women with low platelet counts. Moreover, they have few side-effects and are contraceptive. High-dose intravenous Premarin is also useful but only for a couple of days after which heavy bleeding will ensue. Progestin hormones are similarly effective and are also contraceptive.

Oral contraceptive pills are routinely used to control uterine bleeding in thrombocytopenia secondary to bone marrow failure, chemotherapy and/or stem cell transplantation, during episodes of severe thrombocytopenia. There are no current data supporting whether the use of hormonal management is necessary in addition to platelet transfusion. We expect to show that using continuous OCP in addition to having platelet transfusions will result in a better and more rapid control of uterine bleeding than having platelet transfusions only.

Eligible subjects will be hemodynamically stable, menstruating women aged 12-55, who have bone marrow failure, or are undergoing chemotherapy and/or stem cell transplantation for other diseases with platelet levels less than 50,000/ microliter and present with heavy menstrual bleeding which is expected to last at least 2 weeks. Subjects will be randomized to either continuous OCP (Lo-ovral) 1 tablet twice daily or placebo twice daily for one week. All subjects will receive platelet transfusions to keep platelet levels above 20,000 per microliter throughout the study. After one week, all subjects who continue to bleed will receive continuous OCP 1 tablet twice daily. Those who have stopped bleeding will receive continuous OCP 1 tablet daily. Treatments will be compared for the proportion who stop vaginal bleeding 7 and 14 days after starting treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women aged 12-55 years who have a uterus and at least one functioning ovary.

Women with any active uterine bleeding more than spotting

Diagnosed with bone marrow failure, and other disease that require treatment with chemotherapy or stem cell transplantation with platelet counts less than 50,000 microliters at study entry

Do not desire pregnancy for the duration of the study.

Willing and able to give informed consent.

Willing and able to comply with study requirements.

EXCLUSION CRITERIA:

Age less than 12 years

Postmenopausal women

Hormone level in menopausal range: Follicle Stimulating Hormone greater than 40 IU/L, E (2) less than 20 pg/ml

History of liver disease that precludes OCP use

History of thrombosis, thromboembolism and/or thrombophilia.

Currently on 2 or more tablets of any oral contraceptive pills per day at study entry

Having 2 or more depo medroxyprogesterone acetate injections in the past 12 months or having depo medroxyprogesterone acetate injection in the past 90 days

Leuprolide acetate injection in the past 30 days

Smoker over the age of 35

Women with estrogen dependent tumor e.g. breast cancer.

Pregnancy.

Underlying sickle cell anemia

Women who are taking chemotherapeutic agents known to cause ovarian failure such as alkylating agents

Allergy to any medication in this protocol

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Stratton, MD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amsterdam A, Jakubowski A, Castro-Malaspina H, Baxi E, Kauff N, Krychman M, Stier E, Castiel M. Treatment of menorrhagia in women undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2004 Aug;34(4):363-6. doi: 10.1038/sj.bmt.1704577. PMID 15195079
- [Background] Girling JE, Rogers PA. Recent advances in endometrial angiogenesis research. Angiogenesis. 2005;8(2):89-99. doi: 10.1007/s10456-005-9006-9. Epub 2005 Oct 7. PMID 16211359
- [Background] Fraser IS, Critchley HO, Munro MG, Broder M. Can we achieve international agreement on terminologies and definitions used to describe abnormalities of menstrual bleeding? Hum Reprod. 2007 Mar;22(3):635-43. doi: 10.1093/humrep/del478. Epub 2007 Jan 4. PMID 17204526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lo-ovral | Sugar Pill
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lo-ovral | Sugar Pill | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Categorical [Number; unit: participants]
  <=18 years | 1 |  | 1
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Stop Vaginal Bleeding or Spotting.
Time Frame: 1 week
Population: Early termination because of insufficient accrual. With only one study participant, data could not be analyzed.
Arm/Group | Lo-ovral | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion Who Stop Uterine Bleeding by Day 14.
Time Frame: 2 weeks
Population: Early termination because of insufficient accrual. With only one study participant, data could not be analyzed.
Arm/Group | Lo-ovral | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Total Number of Bleeding Days During the First 7 Days.
Time Frame: 1 week
Population: Early termination because of insufficient accrual. With only one study participant, data could not be analyzed.
Arm/Group | Lo-ovral | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Early termination because of insufficient accrual. With only one study participant, data could not be analyzed. No adverse events data was collected.
Arm/Group | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination because of insufficient accrual. With only one study participant, data could not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes